CLINICAL TRIAL: NCT05690737
Title: A Randomized Controlled Trail to Examine the Efficacy of Tai Chi for the Prophylaxis of Episodic Migraine Compared With Standard Prophylactic Medication in Chinese Women and a Pre-post Neuroimaging and Laboratory-based Study to Explore the Mechanism of Tai Chi's Intervention Effect
Brief Title: Tai Chi for the Prophylaxis of Episodic Migraine: the Efficacy Examination and Mechanism Exploration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, XIE Yao Jie Grace, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A0041948
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Migraine Disorders
Keywords: Migraine; Tai Chi; Women; Mechanism; Prophylaxis
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tai Chi training (Experimental): The participants in this arm will receive 24-week Tai Chi training (1 hour per day, 5 days per week) with 24-week follow-up. A modified 33-short form Yang-style Tai Chi Chuan will be adopted.
  Interventions: Behavioral: Tai Chi training
- Standard prophylactic medication (Active Comparator): Participants in this arm will receive 48-week standard migraine prophylactic medication following neurologist's recommendation.
  Interventions: Drug: Standard prophylactic medication

INTERVENTIONS:
Behavioral: Tai Chi training — The 24-week Tai Chi training will be prescribed with three 1-hour instructor-led sessions and two 1-hour self-practice sessions per week. A modified 33-short form Yang-style Tai Chi Chuan will be adopted. The Tai Chi sessions will be operated by qualified/certified instructors. Each 1-hour training session will consist of 10 minutes brief warm-up stretching session followed by 45 minutes standard Tai Chi routine activities, and 5 minutes of cool-down stretching. The Tai Chi instructors will have to attend a training session that ensure all of them will deliver the same intervention protocol throughout the study. The research assistant will monitor the fidelity of intervention by visiting the Tai Chi sessions frequently. The training activity will be delivered in group. The group size is 25-30 persons. During the 24 weeks follow-up period, the participants are required to practice Tai Chi with the same frequency by themselves.
  Arms: Tai Chi training
Drug: Standard prophylactic medication — Participants assigned to the control group will follow the collaborated neurologist's recommendation, to take the prophylactic medication. The Multidisciplinary Panel on Neuropathic Pain (MPNP) of Hong Kong has published the treatment algorithm for migraine, which is in line with the guideline of the Scottish Intercollegiate Guidelines Network (SIGN) on the pharmacological management of migraine (SIGN 155). Beta-blockers, specifically metoprolol and propranolol, are one of the first-line treatments for migraine prophylaxis. The dosage will start on 10mg and slowly increase by 10mg every week until the dosage reached the highest dose of 150mg/day. The whole course will last for 48 weeks. The second line drug such as amitriptyline and the third line drug such as gabapentin will be adopted according to doctor's judgement if necessary. RA will help the participants to make appointment with the neurological doctor, to obtain the prescription. The adverse events will be recorded accordingly.
  Arms: Standard prophylactic medication

SUMMARY:
The proposed study aims to examine the clinical efficacy of 24-week Tai Chi training in the prophylaxis of episodic migraine comparing with standard prophylactic medication in Hong Kong Chinese women, and to explore the mechanism of Tai Chi's intervention effect by examining the associations of changes in migraine features with neurovascular and neuroinflammation variations.

DETAILED DESCRIPTION:
A two-arm individual level randomized controlled trial is designed. A total of 220 local women diagnosed with episodic migraine between 18-65 years will be randomly assigned to one of two groups: 1) a Tai Chi training group receiving the 33-short form Yang-style Tai Chi training; or 2) a standard prophylactic medication group receiving the regular medication prescribed by the neurologist. The intervention period will be 24 weeks with another 24 weeks follow-up. The frequency of migraine attack, migraine days, intensity and duration of headache will be recorded by a migraine diary at the baseline, 24th weeks, and 48th weeks. Other outcomes including migraine related disability, stress, sleep quality, fatigue, and QOL will be measured at these three time points. The clinical efficacy will be determined by comparing the differences of outcomes from baseline to the end of the trial between two groups. The MRI and TCD will be used to measure the degree of white matter abnormality and cerebrovascular function, respectively; and the inflammatory markers will also be tested at three time points for Tai Chi participants. The mechanism of intervention effect will be explored by analyzing the changes and associations of migraine features with the process of these neurovascular functions and inflammatory markers during and after the Tai Chi training.

ELIGIBILITY:
Inclusion Criteria:

* Chinese woman, aged 18-65 years.
* Have a clinical diagnosis of episodic migraine (migraine with less than 15 attacks per month) with or without aura according to the International Classification of Headache Disorders, 3rd edition (ICHD-3).
* First migraine attack before the age of 45 years.
* Between two and six migraine attacks in one month.
* At least one of the following migraine characteristics is met: nausea, vomiting, photophobia, or phonophobia.
* Duration of migraine attacks is 2-72 h without acute medication or at least 1 h with acute medication.
* Able to undertake designated level of Tai Chi exercise.
* Live in Hong Kong.

Exclusion Criteria:

* Severe migraine attacks with disabilities that cannot perform moderate intensity physical activity.
* Secondary headache and other neurological disease.
* More than 5 days of non-migrainous headache per month.
* Experience with Tai Chi or other body-mind exercises (yoga, biofeedback, medication, etc.) after diagnosis of migraine.
* Undergoing other alternative therapeutic treatments during recruitment period, or received other alternative therapeutic treatments in the past 12 weeks.
* Pregnancy, lactation period, or currently using contraceptives.
* Use of pharmacological prophylactic treatment for migraine in the past 12 weeks.
* Drug abuse, take antipsychotic or antidepressant drugs, or take analgesics for other chronic pain more than 3 days a month in the past 12 weeks.
* Epilepsy, or have a psychiatric disease.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference in frequency of migraine attacks | Between 4 weeks before randomization and weeks 21-24 / 45-48 after randomization
  The frequency of migraine attacks will be measured by the number of attacks per month.
The difference in frequency of migraine days | Between 4 weeks before randomization and weeks 21-24 / 45-48 after randomization
  The frequency of migraine days will be measured by the days with migraine attacks per month.
The difference of white matter abnormalities (WMAs) | From the baseline to 24 weeks and 48 weeks
  All the participants in the Tai Chi group will be measured with MRI. The appearance, number, size and location of WMAs will be recorded. Two experienced neurologists or neuroradiologists will be invited to review the MRI scans independently. Scheltens' visual rating scale will be used to measure the degree of WMAs. Briefly, WMAs will be separately graded in each of the following locations: frontal lobes, temporal lobes, parietal lobes and occipital lobes. WMAs will be graded as follows: 0 (no lesions), 1 (hyperintensity < 3 mm and n ≤ 5), 2 (< 3 mm and n ≥ 6), 3 (4-10 mm and n ≤ 5), 4 (4-10 mm and n ≥ 6), 5 (≥ 11 mm and n ≥ 1), and 6 (confluent). The sum of scores from each location will be considered as the final score. Only the women who are identified WMAs (Scheltens' visual rating scores >0) will take the MRI test again at the 24th week and 48th week.
The difference of pulsatility index (PI) | From the baseline to 24 weeks and 48 weeks
  PI in all intracranial and neck vessels will be measured and recorded by Transcranial Doppler (TCD).
The difference of mean blood flow velocity (MBFV) | From the baseline to 24 weeks and 48 weeks
  MBFV in all intracranial and neck vessels will be measured and recorded by Transcranial Doppler (TCD).
The difference of impaired cerebrovascular responsiveness (CVR). | From the baseline to 24 weeks and 48 weeks
  The CVR will be calculated by: CVR=△MBFV=(Vstim-Vrest)/Vrest*100, where △MBFV is the relative change of blood flow velocity, Vstim is the blood flow velocity during the stimulation, and Vrest is the baseline flow velocity during the initial 5 min prior to stimulation. The value will be calculated by the mean of both left and right brain and from 10 cycles.

SECONDARY OUTCOMES:
The proportion of responders | Between 4 weeks before randomization and weeks 21-24 / 45-48 after randomization
  Defined as the proportion of patients with at least a 50% reduction of the number of attacks per month
The intensity of the headache | Between 4 weeks before randomization and weeks 21-24 / 45-48 after randomization
  The intensity of the headache measured by a Visual Analogue Scale (VAS). This scale is most commonly anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 10). Higher scores indicate higher level of headache intensity.
The duration of headache | Between 4 weeks before randomization and weeks 21-24 / 45-48 after randomization
  The duration of headache recorded in the migraine diary to the nearest 0.1 hour.
Migraine related disability | From the baseline to 24 weeks and 48 weeks
  Migraine related disability measured by the Migraine Disability Assessment Score (MIDAS). The MIDAS consists of five items that reflect the number of days reported as either missing or with reduced productivity at work, home, and social events in last 3 months and two additional items that assess the number of days with headaches in the last 3 months and a scale of the painfulness of the headaches. The MIDAS is scored as the sum of days reported in the first five questions. Higher scores are indicative of more disability.
Stress level | From the baseline to 24 weeks and 48 weeks
  Stress level evaluated by the Perceived Stress Scale-14 (PSS-14). The total score of PSS-14 ranges from 0 to 56 with higher scores indicating higher perceived stress.
Sleep quality | From the baseline to 24 weeks and 48 weeks
  Sleep quality examined by the Chinese version of the Pittsburgh Sleep Quality Index (PSQI). The global score of PSQI ranges from 0 to 21 with a higher score indicating worse sleep quality.
Fatigue level | From the baseline to 24 weeks and 48 weeks
  Fatigue level evaluated by the Numeric Rating Scale-fatigue scale (NRS). NRS evaluates fatigue level at a 0-to-10 scale, with 0 indicating no fatigue and 10 indicating the worst possible fatigue.
Health related Quality-of-Life | From the baseline to 24 weeks and 48 weeks
  Health related Quality-of-Life measured by the Migraine-Specific Quality-of-Life Questionnaire (MSQ). The total scores of MSQ range from 0-100, with a higher score indicating better Quality-of-Life.
Weight | From the baseline to 24 weeks and 48 weeks
  Weight in kilograms
Height | From the baseline to 24 weeks and 48 weeks
  Height in meters
Waist circumference | From the baseline to 24 weeks and 48 weeks
  Waist circumference in cm
Hip circumference | From the baseline to 24 weeks and 48 weeks
  Hip circumference in cm
Percent body fat | From the baseline to 24 weeks and 48 weeks
  Percent body fat in %
TNF- α | From the baseline to 24 weeks and 48 weeks
  The blood samples (10 ml) will be drawn from antecubital vein of all eligible participants by a research nurse. Serum is separated after centrifugation for 10 minutes at 2,000g and frozen at - 20 °C until assay. The serum sample will be sent to medical laboratories for testing by the Enzyme-linked immunosorbent assay (ELISA). TNF-α will be measured in pg/ml.
CGRP | From the baseline to 24 weeks and 48 weeks
  The blood samples (10 ml) will be drawn from antecubital vein of all eligible participants by a research nurse. Serum is separated after centrifugation for 10 minutes at 2,000g and frozen at - 20 °C until assay. The serum sample will be sent to medical laboratories for testing by the Enzyme-linked immunosorbent assay (ELISA). CGRP will be measured in pg/ml.
CRP | From the baseline to 24 weeks and 48 weeks
  The blood samples (10 ml) will be drawn from antecubital vein of all eligible participants by a research nurse. Serum is separated after centrifugation for 10 minutes at 2,000g and frozen at - 20 °C until assay. The serum sample will be sent to medical laboratories for testing by the Enzyme-linked immunosorbent assay (ELISA). CRP will be measured in pg/ml.
IL-6 | From the baseline to 24 weeks and 48 weeks
  The blood samples (10 ml) will be drawn from antecubital vein of all eligible participants by a research nurse. Serum is separated after centrifugation for 10 minutes at 2,000g and frozen at - 20 °C until assay. The serum sample will be sent to medical laboratories for testing by the Enzyme-linked immunosorbent assay (ELISA). IL-6 will be measured in pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Jie Xie, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - The Hong Kong Polytechnic University, Hong Kong, HONG KONG
  - The Hong Kong Polytechnic University, Hung Hom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xie YJ, Liao X, Hui SS, Tian L, Yeung WF, Lau AY, Tyrovolas S, Gao Y, Chen X. Tai Chi for the prophylaxis of episodic migraine: protocol of a non-inferiority randomized controlled trial with mechanism exploration. BMC Complement Med Ther. 2023 Sep 18;23(1):328. doi: 10.1186/s12906-023-04154-x. PMID 37723467